CLINICAL TRIAL: NCT00001772
Title: Evaluation of Patients With Rapid Cycling Bipolar Disorder
Brief Title: Evaluation of Patients With Rapid Cycling Bipolar Disorder (RCBD)
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980156; 98-M-0156
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-08

CONDITIONS: Bipolar Disorder; Rapid Cycling Bipolar Disorder
Keywords: Bipolar Disorder; Rapid Cycling; Screening
MeSH Terms: conditions — Bipolar Disorder

SUMMARY:
Bipolar disorder is a mood (affective) disorder characterized by the occurrence of alternating feelings of excitement (mania) and depression. It is a common, but serious condition, and potentially life-threatening. Patients are considered to have a rapid cycling form of bipolar disorder if they experience four or more episodes of hypomania (mild degree of mania), mania, and/or depression. Approximately 20% of the patients in bipolar clinics have the rapid cycling form of the disorder. Therefore it can be said that RCBD is not a rare condition and that it can severely impair a patient. These reasons alone justify studying RCBD. However, researchers also believe that information gathered by studying patients with RCBD can be used while studying other patients with different forms of bipolar disorder.

The purpose of this study is to screen patients diagnosed as having rapid cycling bipolar disorder to see if they fit the criteria for the diagnosis and to see if they would be interested in participating in other research studies.

Patients will undergo diagnostic interviews, physical examination, routine blood tests, EKG (electrocardiogram), and complete self-rating forms as part of the screening process.

DETAILED DESCRIPTION:
The purpose of this protocol is to allow for the medical and psychiatric screening of patients with rapid cycling bipolar disorder in order to ascertain (1) that they fit the criteria for the diagnosis; and (2) that they are interested in participating in one of our research projects. Patients will undergo diagnostic interviews, complete self-rating forms, and have a physical examination, routine blood tests, and an electrocardiogram.

ELIGIBILITY:
Must be currently in treatment with a psychiatrist.

Subjects must not have borderline or antisocial personality disorders, must not meet criteria for substance abuse or dependence within the past six months.

Subjects must not have significant hepatic, renal, endocrine, or cardiovascular disease.

Subjects must not be pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1998-09; Study Completion 2001-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Dunner DL, Fieve RR. Clinical factors in lithium carbonate prophylaxis failure. Arch Gen Psychiatry. 1974 Feb;30(2):229-33. doi: 10.1001/archpsyc.1974.01760080077013. No abstract available. PMID 4589148
- [Background] Coryell W, Endicott J, Keller M. Rapidly cycling affective disorder. Demographics, diagnosis, family history, and course. Arch Gen Psychiatry. 1992 Feb;49(2):126-31. doi: 10.1001/archpsyc.1992.01820020046006. PMID 1550465
- [Background] Leibenluft E. Women with bipolar illness: clinical and research issues. Am J Psychiatry. 1996 Feb;153(2):163-73. doi: 10.1176/ajp.153.2.163. PMID 8561195